CLINICAL TRIAL: NCT01236794
Title: Community-Based Participatory Research to Improve Health and Quality of Life of Latino Youth: Every Little Step Counts
Acronym: ELSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); St. Vincent de Paul Medical and Dental Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P20MD002316ELSC; P20MD002316 (NIH)
Record Dates: First submitted 2010-09-14; First posted 2010-11-09 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2018-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle and Exercise Intervention (Experimental)
  Interventions: Behavioral: Lifestyle Education Sessions and Youth Exercise Sessions

INTERVENTIONS:
Behavioral: Lifestyle Education Sessions and Youth Exercise Sessions — The intervention will include a ~1-2 hour weekly education session to address the following constructs: health awareness, healthy eating, physical activity, roles and responsibilities, self-esteem, self-efficacy, diabetes knowledge, communication, and peer / family relationships. In addition to the education classes youth will participate in 3 exercise sessions per week (~1-1.5 hrs) that will consist of individual and group physical activities to include both aerobic and resistance exercises. The exercise intensity will progressively increase over the 12-week intervention. Both the education and activity sessions will be delivered at the Lincoln Family YMCA.
  Other Names: ELSC; Every Little Step Counts

SUMMARY:
The purpose of this study is to examine the effects of a lifestyle intervention program on type 2 diabetes risk factors and quality of life in overweight Latino youth.

DETAILED DESCRIPTION:
With the increasing prevalence of obesity, the incidence of obesity-related co-morbidities including depression and type 2 diabetes have emerged as critical public health conditions. Furthermore, Latinos experience a disproportionately greater burden of these obesity-related disorders. Therefore, we have developed a 12-week community-based lifestyle intervention that includes weekly education sessions for children and their parents and 3 exercise sessions per week for youth. The program will be delivered at a local YMCA in the greater Phoenix Metropolitan area.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic Ethnicity (Child and Parent)
* Age 14-16 (Child) and Parent age < 85
* BMI Percentile above the 85th (child)
* Ability to read and speak English (child)

Exclusion Criteria:

* Taking medication(s) or diagnosed with a condition that could influence exercise ability or carbohydrate metabolism (e.g., polycystic ovarian syndrome, exercise induced asthma, orthopedic limitations) (Child and (Parent OGTT only))
* Involved in any formal weight-loss program in the past 6 months (Child)
* Diagnosed diabetes (type 1 or type 2 Child)
* Weight is less than 110 Ibs (Child and Parent)

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity | About 12 Weeks
  Insulin sensitivity will be determined using a insulin and glucose values collected during a 2-hour oral glucose tolerance test.

SECONDARY OUTCOMES:
QOL | About 12 Weeks
  Weight-specific quality of Life will be determined by self report using a multicultural quality of life instrument for adolescents

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shaibi GQ, Konopken Y, Hoppin E, Keller CS, Ortega R, Castro FG. Effects of a culturally grounded community-based diabetes prevention program for obese Latino adolescents. Diabetes Educ. 2012 Jul-Aug;38(4):504-12. doi: 10.1177/0145721712446635. Epub 2012 May 14. PMID 22585870
- [Result] Shaibi GQ, Greenwood-Ericksen MB, Chapman CR, Konopken Y, Ertl J. Development, implementation, and effects of community-based diabetes prevention program for obese latino youth. J Prim Care Community Health. 2010 Oct 1;1(3):206-12. doi: 10.1177/2150131910377909. PMID 21461141
- [Result] Ryder JR, Vega-Lopez S, Ortega R, Konopken Y, Shaibi GQ. Lifestyle intervention improves lipoprotein particle size and distribution without weight loss in obese Latino adolescents. Pediatr Obes. 2013 Oct;8(5):e59-63. doi: 10.1111/j.2047-6310.2013.00162.x. Epub 2013 Apr 10. PMID 23576420